CLINICAL TRIAL: NCT01064687
Title: A Randomized, Placebo-Controlled Comparison of the Effects of Two Doses of LY2189265 or Exenatide on Glycemic Control in Patients With Type 2 Diabetes on Stable Doses of Metformin and Pioglitazone (AWARD-1: Assessment of Weekly Administration of LY2189265 in Diabetes-1)
Brief Title: A Study in Participants With Type 2 Diabetes Mellitus
Acronym: AWARD-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11373; H9X-MC-GBDA (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide; Exenatide; Metformin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1.5 mg LY2189265 (Experimental): LY2189265 (Dulaglutide): 1.5 milligrams (mg), subcutaneous (SC), once weekly for 52 weeks
  Metformin: at least 1500 milligrams per day (mg/day), oral, for 52 weeks
  Pioglitazone: at least 30 mg/day, oral, for 52 weeks
  Interventions: Drug: LY2189265; Drug: Metformin; Drug: Pioglitazone
- 0.75 mg LY2189265 (Experimental): LY2189265 (Dulaglutide): 0.75 milligrams (mg), subcutaneous (SC), once weekly for 52 weeks
  Metformin: at least 1500 milligrams per day (mg/day), oral, for 52 weeks
  Pioglitazone: at least 30 mg/day, oral, for 52 weeks
  Interventions: Drug: LY2189265; Drug: Metformin; Drug: Pioglitazone
- Exenatide (Active Comparator): Exenatide: 5 micrograms (mcg), subcutaneous (SC), twice daily for 4 weeks, followed by 10 mcg, SC, twice daily for 48 weeks
  Metformin: at least 1500 milligrams per day (mg/day), oral, for 52 weeks
  Pioglitazone: at least 30 mg/day, oral, for 52 weeks
  Interventions: Drug: Exenatide; Drug: Metformin; Drug: Pioglitazone
- Placebo (Placebo Comparator): Placebo: subcutaneous (SC), once weekly for 26 weeks
  LY2189265 (Dulaglutide): After 26 weeks, participants were randomized to receive either 0.75 milligrams (mg) or 1.5 mg, SC, once weekly for an additional 26 weeks (from week 26 through week 52).
  Metformin: at least 1500 milligrams per day (mg/day), oral, for 52 weeks
  Pioglitazone: at least 30 mg/day, oral, for 52 weeks
  Interventions: Drug: LY2189265; Drug: Placebo; Drug: Metformin; Drug: Pioglitazone

INTERVENTIONS:
Drug: LY2189265
  Other Names: Dulaglutide
  Arms: 0.75 mg LY2189265; 1.5 mg LY2189265; Placebo
Drug: Exenatide
  Arms: Exenatide
Drug: Placebo
  Arms: Placebo
Drug: Metformin
Drug: Pioglitazone

SUMMARY:
The purpose of this study is to determine if LY2189265 is effective and safe in reducing hemoglobin A1c (HbA1c), as compared to placebo (no medicine), or exenatide in participants with Type 2 Diabetes. The participants must also be taking metformin and pioglitazone.

DETAILED DESCRIPTION:
During the study, if a participant developed persistent, severe hyperglycemia despite full compliance with the assigned therapeutic regimen, the participant received additional therapeutic intervention or initiation of an alternative antihyperglycemic medication following study drug discontinuation (rescue therapy). Participants who received rescue therapy were included in the analysis population, but only measurements obtained prior to the beginning of rescue therapy were included in specified analyses.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes (T2D) not well controlled on 1, 2, or 3 oral antidiabetic medications

  1. Glycosylated hemoglobin (HbA1c) greater than or equal to 7 and less than or equal to 11 if taking 1 oral antidiabetic medication
  2. HbA1c greater than or equal to 7 and less than or equal to 10 if on 2 or 3 oral antidiabetic medications
* Able to tolerate minimum dose of 1500 milligrams (mg) metformin a day and 30 mg pioglitazone per day.
* Willing to inject subcutaneous (SC) medication up to 2 times per day
* Stable weight for 3 months prior to screening
* Body mass index (BMI) between 23 and 45 kilograms per meter squared (kg/m^2)
* Females of child bearing potential must test negative for pregnancy at screening by serum pregnancy test and be willing to use a reliable method of birth control during the study and for 1 month following the last dose of study drug.

Exclusion Criteria:

* Type 1 Diabetes
* HbA1c equal to or less than 6.5 before randomization or at randomization
* Chronic insulin use
* Taking drugs to promote weight loss by prescription or over the counter
* Taking systemic steroids for greater than 14 days except for topical, eye, nasal, or inhaled
* History of fluid retention or edema
* History of Heart Failure New York Heart Classification II, III, or IV or acute myocardial infarction or stroke within 2 months of screening
* Gastrointestinal (GI; stomach) problems such as diabetic gastroparesis or bariatric surgery (stomach stapling) or chronically taking drugs that directly affect GI motility
* Hepatitis or liver disease or alanine transaminase (ALT) greater than 2.5 times the upper limit of normal
* Acute or chronic pancreatitis of any form
* Renal disease (kidney) with a serum creatinine of greater than or equal to 1.5 milligrams per deciliter (mg/dL) for males and greater than or equal to 1.4 mg/dL for females, or a creatine clearance of less than 60 milliliters per minute (mL/min)
* History (includes family) of type 2A or 2B Multiple Endocrine Neoplasia (MEN 2A or 2B) or medullary c-cell hyperplasia or thyroid cancer
* A serum calcitonin greater than or equal to 20 picograms per milliliter (pg/mL) at screening
* Significant active autoimmune disease such as Lupus or Rheumatoid Arthritis
* History of or active malignancy except skin or in situ cervical or prostate cancer for within last 5 years
* Sickle cell, hemolytic anemia, or other hematological condition that may interfere with HbA1c testing
* Organ transplant except cornea
* Have enrolled in another clinical trial within the last 30 days
* Have previously signed an informed consent or participated in a LY2189265 (dulaglutide) study
* Have taken a glucagon-like peptide 1 (GLP-1) receptor agonist within the 3 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 978 (Actual)
Dates: Start 2010-02; Primary Completion 2011-11 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (89):
- United States (78):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goodyear, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cathedral City, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fresno, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenbrae, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lancaster, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mission Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterey, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., National City, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oceanside, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paramount, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roseville, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Ramon, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tustin, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Britain, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hollywood, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pembroke Pines, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boise, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Meridian, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Crystal Lake, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vincennes, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madisonville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Orleans, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangor, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Biddeford, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elkridge, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bloomfield Hills, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Flint, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashua, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albany, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Flushing, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Syracuse, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Asheville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cary, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morehead City, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbus, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dayton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Delaware, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Perrysburg, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bend, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Corvallis, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eugene, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beaver, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danville, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Levittown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wilkes-Barre, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greer, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Myrtle Beach, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arlington, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Corpus Christi, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., El Paso, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Schertz, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ogden, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. George, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Jordan, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tacoma, Washington
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires, Argentina
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- Puerto Rico (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caguas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hato Rey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manatí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Germán
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yabucoa

REFERENCES:
- [Derived] Ferdinand KC, Dunn J, Nicolay C, Sam F, Blue EK, Wang H. Weight-dependent and weight-independent effects of dulaglutide on blood pressure in patients with type 2 diabetes. Cardiovasc Diabetol. 2023 Mar 9;22(1):49. doi: 10.1186/s12933-023-01775-x. PMID 36894938
- [Derived] Boustani MA, Pittman I 4th, Yu M, Thieu VT, Varnado OJ, Juneja R. Similar efficacy and safety of once-weekly dulaglutide in patients with type 2 diabetes aged >/=65 and <65 years. Diabetes Obes Metab. 2016 Aug;18(8):820-8. doi: 10.1111/dom.12687. Epub 2016 Jun 7. PMID 27161178
- [Derived] Yu M, Van Brunt K, Varnado OJ, Boye KS. Patient-reported outcome results in patients with type 2 diabetes treated with once-weekly dulaglutide: data from the AWARD phase III clinical trial programme. Diabetes Obes Metab. 2016 Apr;18(4):419-24. doi: 10.1111/dom.12624. Epub 2016 Feb 4. PMID 26691396

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to ethical considerations and to preserve the blinding of the study, participants randomized to placebo at baseline were reassigned at 26 weeks to either 1.5 mg LY2189265 or 0.75 mg LY2189265 from 26 weeks through 52 weeks.
Groups:
- Placebo: Placebo: subcutaneous (SC), once weekly for 26 weeks
  Metformin: at least 1500 milligrams per day (mg/day), oral, for 26 weeks
  Pioglitazone: at least 30 mg/day, oral, for 26 weeks
Period: Overall Study
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Started | 279 | 280 | 278 (Of 278 participants randomized to Exenatide, 2 chose not to take study drug.) | 141
Received at Least 1 Dose of Study Drug | 279 | 280 | 276 | 141
Completed 26 Weeks | 260 | 263 | 252 | 124
Completed | 245 | 254 | 237 | 124
Not Completed | 34 | 26 | 41 | 17
Not completed — Adverse Event | 9 | 4 | 10 | 3
Not completed — Death | 1 | 1 | 0 | 0
Not completed — Entry Criteria Not Met | 3 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 2 | 3
Not completed — Lost to Follow-up | 7 | 10 | 13 | 5
Not completed — Physician Decision | 2 | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 1
Not completed — Sponsor Decision | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 9 | 7 | 12 | 5
Not completed — Treatment Noncompliance | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who were randomized and received at least 1 dose of LY2189265, Exenatide, or Placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo | Total
Number analyzed (Participants) | 279 | 280 | 276 | 141 | 976
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.25 (9.72) | 55.79 (9.45) | 55.45 (10.15) | 54.56 (10.01) | 55.65 (9.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 112 | 120 | 58 | 406
  Male | 163 | 168 | 156 | 83 | 570
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 93 | 102 | 91 | 45 | 331
  Not Hispanic or Latino | 186 | 178 | 184 | 96 | 644
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 40 | 37 | 38 | 20 | 135
  Asian | 6 | 8 | 4 | 6 | 24
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 0 | 3
  Black or African American | 24 | 24 | 18 | 10 | 76
  White | 205 | 207 | 211 | 103 | 726
  More than one race | 3 | 3 | 3 | 2 | 11
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 226 | 226 | 223 | 113 | 788
  Mexico | 37 | 36 | 35 | 19 | 127
  Argentina | 16 | 18 | 18 | 9 | 61
Body Weight [Mean (Standard Deviation); unit: kilograms] | 96.22 (19.63) | 95.53 (20.56) | 97.37 (18.87) | 94.12 (19.28) | 96.04 (19.64)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter squared (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms per meter squared (kg/m^2) | 33.09 (5.33) | 33.00 (5.50) | 33.54 (5.36) | 32.90 (5.66) | 33.16 (5.43)
Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 8.10 (1.34) | 8.05 (1.24) | 8.07 (1.34) | 8.06 (1.31) | 8.07 (1.31)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 8.76 (5.59) | 8.78 (5.47) | 8.84 (5.71) | 8.60 (5.78) | 8.76 (5.61)
Fasting Serum Glucose [Mean (Standard Deviation); unit: millimoles per liter (mmol/L)] | 9.00 (3.09) | 8.84 (2.76) | 9.11 (3.04) | 9.22 (3.01) | 9.02 (2.97)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 26 Weeks Endpoint in Glycosylated Hemoglobin (HbA1c)
Description: Least squares (LS) means were calculated using analysis of covariance (ANCOVA) with country and treatment as fixed effects and baseline HbA1c as a covariate.
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265, Exenatide, or Placebo with evaluable HbA1c data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 271 | 269 | 266 | 119
percentage of glycosylated hemoglobin | -1.51 (0.06) | -1.30 (0.06) | -0.99 (0.06) | -0.46 (0.08)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Placebo; Superiority analysis; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is adjusted for multiplicity based on a tree-gatekeeping strategy. To determine significance, p-value is compared to the family-wise 1-sided Type I error of 0.025. The confidence interval is not adjusted for multiplicity; LS Mean Difference = -1.05, 95% CI 2-sided [-1.22 to -0.88]
Statistical Analysis 2: Comparison: 1.5 mg LY2189265 vs Exenatide; Non-inferiority analysis; Test type: Non-Inferiority or Equivalence — A non-inferiority margin of 0.4% was used; p < 0.0001, ANCOVA — P-value is adjusted for multiplicity, based on tree-gatekeeping strategy. To determine significance, p-value is compared to the family-wise 1-sided Type I error of 0.025. The confidence interval is not adjusted for multiplicity; LS Mean Difference = -0.52, 95% CI 2-sided [-0.66 to -0.39]
Statistical Analysis 3: Comparison: 0.75 mg LY2189265 vs Placebo; Superiority analysis; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.84, 95% CI 2-sided [-1.01 to -0.67]
Statistical Analysis 4: Comparison: 1.5 mg LY2189265 vs Exenatide; Superiority analysis; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.52, 95% CI 2-sided [-0.66 to -0.39]
Statistical Analysis 5: Comparison: 0.75 mg LY2189265 vs Exenatide; Non-inferiority analysis; Test type: Non-Inferiority or Equivalence — A non-inferiority margin of 0.4% was used; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.31, 95% CI 2-sided [-0.44 to -0.18]
Statistical Analysis 6: Comparison: 0.75 mg LY2189265 vs Exenatide; Superiority analysis; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.31, 95% CI 2-sided [-0.44 to -0.18]

2. Secondary Outcome: Change From Baseline to 52 Weeks Endpoint in Glycosylated Hemoglobin (HbA1c)
Description: as for outcome 1
Time Frame: Baseline, 52 weeks
Population: Participants who were randomized at baseline to LY2189265 or Exenatide and received at least 1 dose of study drug with evaluable HbA1c data. Only pre-rescue measurements were used. LOCF was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide
Number analyzed (Participants) | 271 | 269 | 266
percentage of glycosylated hemoglobin | -1.36 (0.08) | -1.07 (0.08) | -0.80 (0.08)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Exenatide; Non-inferiority analysis; Test type: Non-Inferiority or Equivalence — A non-inferiority margin of 0.4% was used; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.56, 95% CI 2-sided [-0.73 to -0.39]
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Exenatide; Non-inferiority analysis; Test type: Non-Inferiority or Equivalence — A non-inferiority margin of 0.4% was used; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.27, 95% CI 2-sided [-0.44 to -0.11]
Statistical Analysis 3: Comparison: 1.5 mg LY2189265 vs Exenatide; Superiority analysis; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.56, 95% CI 2-sided [-0.73 to -0.39]
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Exenatide; Superiority analysis; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS Mean Difference = -0.27, 95% CI 2-sided [-0.44 to -0.11]

3. Secondary Outcome: Change From Baseline to 26 Weeks for Body Weight
Description: Least squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) analysis with treatment, country, visit, and treatment-by-visit as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265, Exenatide, or Placebo with evaluable body weight data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 259 | 253 | 245 | 109
kilograms (kg) | -1.34 (0.25) | 0.18 (0.25) | -1.14 (0.26) | 1.37 (0.37)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -2.72, 95% CI 2-sided [-3.58 to -1.85]
Statistical Analysis 2: Comparison: 1.5 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p = 0.571, Mixed Models Analysis; LS Mean Difference = -0.20, 95% CI 2-sided [-0.88 to 0.49]
Statistical Analysis 3: Comparison: 0.75 mg LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis; LS Mean Difference = -1.19, 95% CI 2-sided [-2.06 to -0.33]
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = 1.33, 95% CI 2-sided [0.64 to 2.01]
Statistical Analysis 5: Comparison: Exenatide vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -2.52, 95% CI 2-sided [-3.39 to -1.65]

4. Secondary Outcome: Change From Baseline to 52 Weeks for Body Weight
Description: as for outcome 3
Time Frame: Baseline, 52 weeks
Population: Participants who were randomized at baseline to LY2189265 or Exenatide and received at least 1 dose of study drug with evaluable body weight data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide
Number analyzed (Participants) | 238 | 231 | 210
kilograms (kg) | -1.08 (0.34) | 0.49 (0.34) | -0.76 (0.35)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p = 0.507, Mixed Models Analysis; LS Mean Difference = -0.32, 95% CI 2-sided [-1.25 to 0.62]
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p = 0.009, Mixed Models Analysis; LS Mean Difference = 1.25, 95% CI 2-sided [0.32 to 2.19]

5. Secondary Outcome: Change From Baseline to 26 Weeks on Body Mass Index (BMI)
Description: Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265, Exenatide, or Placebo with evaluable BMI data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: kilograms per meter squared (kg/m^2)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 259 | 253 | 245 | 109
kilograms per meter squared (kg/m^2) | -0.48 (0.09) | 0.07 (0.09) | -0.41 (0.09) | 0.49 (0.13)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Means Difference = -0.97, 95% CI 2-sided [-1.27 to -0.67]
Statistical Analysis 2: Comparison: 1.5 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p = 0.568, Mixed Models Analysis; LS Mean Difference = -0.07, 95% CI 2-sided [-0.31 to 0.17]
Statistical Analysis 3: Comparison: 0.75 mg LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; LS Mean Difference = -0.42, 95% CI 2-sided [-0.72 to -0.12]
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = 0.48, 95% CI 2-sided [0.24 to 0.71]
Statistical Analysis 5: Comparison: Exenatide vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.90, 95% CI 2-sided [-1.20 to -0.60]

6. Secondary Outcome: Change From Baseline to 52 Weeks on Body Mass Index (BMI)
Description: as for outcome 5
Time Frame: Baseline, 52 weeks
Population: Participants who were randomized at baseline to LY2189265 or Exenatide and received at least 1 dose of study drug with evaluable BMI data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: kilograms per meter squared (kg/m^2)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide
Number analyzed (Participants) | 238 | 231 | 210
kilograms per meter squared (kg/m^2) | -0.37 (0.12) | 0.18 (0.12) | -0.28 (0.12)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p = 0.580, Mixed Models Analysis; LS Mean Difference = -0.09, 95% CI 2-sided [-0.42 to 0.23]
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; LS Mean Difference = 0.46, 95% CI 2-sided [0.14 to 0.79]

7. Secondary Outcome: Change From Baseline to 26 Weeks for Daily Mean Blood Glucose Values From the 8-point Self-monitored Plasma Glucose (SMPG) Profiles
Description: The SMPG data were collected at the following 8 time points: pre-morning meal; 2 hours post-morning meal; pre-midday meal; 2 hours post-midday meal; pre-evening; 2 hours post-evening meal; bedtime; and 3AM or 5 hours after bedtime. Least squares (LS) means of the mean of the 8 time points (daily mean) were calculated using a mixed-effects model for repeated measures (MMRM) analysis with treatment, country, visit, and treatment-by-visit as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265, Exenatide, or Placebo with evaluable SMPG data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 207 | 195 | 202 | 78
milligrams per deciliter (mg/dL) | -46.82 (1.81) | -42.09 (1.87) | -37.48 (1.83) | -18.07 (2.68)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -28.76, 95% CI 2-sided [-34.50 to -23.02]
Statistical Analysis 2: Comparison: 1.5 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -9.34, 95% CI 2-sided [-13.62 to -5.06]
Statistical Analysis 3: Comparison: 0.75 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -24.02, 95% CI 2-sided [-29.80 to -18.24]
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p = 0.038, Mixed Models Analysis; LS Mean Difference = -4.61, 95% CI 2-sided [-8.95 to -0.27]
Statistical Analysis 5: Comparison: Exenatide vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -19.41, 95% CI 2-sided [-25.18 to -13.65]

8. Secondary Outcome: Change From Baseline to 52 Weeks for Daily Mean Blood Glucose Values From the 8-point Self-monitored Plasma Glucose (SMPG) Profiles
Description: as for outcome 7
Time Frame: Baseline, 52 weeks
Population: Participants who were randomized at baseline to LY2189265 or Exenatide and received at least 1 dose of study drug with evaluable SMPG data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide
Number analyzed (Participants) | 187 | 185 | 178
milligrams per deciliter (mg/dL) | -43.84 (2.07) | -40.62 (2.12) | -36.16 (2.11)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; LS Mean Difference = -7.68, 95% CI 2-sided [-12.84 to -2.52]
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p = 0.092, Mixed Models Analysis; LS Mean Difference = -4.47, 95% CI 2-sided [-9.66 to 0.73]

9. Secondary Outcome: Percentage of Participants Attaining Glycosylated Hemoglobin (HbA1c) Less Than 7% and Less Than or Equal to 6.5% at 26 Weeks
Description: The percentage of participants achieving HbA1c level less than 7.0% and less than or equal to 6.5% was analyzed with a logistic regression model with baseline, country, and treatment as factors included in the model.
Time Frame: Baseline, 26 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 271 | 269 | 266 | 119
percentage of participants
  HbA1c Less Than 7% | 78.2 | 65.8 | 52.3 | 42.9
  HbA1c Less Than or Equal to 6.5% | 62.7 | 53.2 | 38.0 | 24.4
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison for HbA1c less than 7.0%; Odds Ratio (OR) = 13.1, 95% CI 2-sided [7.4 to 23.4]
Statistical Analysis 2: Comparison: 1.5 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison for HbA1c less than 7.0%; Odds Ratio (OR) = 6.2, 95% CI 2-sided [3.9 to 10.1]
Statistical Analysis 3: Comparison: 0.75 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison for HbA1c less than 7.0%; Odds Ratio (OR) = 4.8, 95% CI 2-sided [2.8 to 8.0]
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison for HbA1c less than 7.0%; Odds Ratio (OR) = 2.3, 95% CI 2-sided [1.5 to 3.5]
Statistical Analysis 5: Comparison: Exenatide vs Placebo; Test type: Superiority or Other; p = 0.004, Regression, Logistic — Treatment comparison for HbA1c less than 7.0%; Odds Ratio (OR) = 2.1, 95% CI 2-sided [1.3 to 3.5]
Statistical Analysis 6: Comparison: 1.5 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison for HbA1c less than or equal to 6.5%; Odds Ratio (OR) = 11.8, 95% CI 2-sided [6.7 to 20.8]
Statistical Analysis 7: Comparison: 1.5 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison for HbA1c less than or equal to 6.5%; Odds Ratio (OR) = 4.4, 95% CI 2-sided [2.9 to 6.8]
Statistical Analysis 8: Comparison: 0.75 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison for HbA1c less than or equal to 6.5%; Odds Ratio (OR) = 6.3, 95% CI 2-sided [3.7 to 10.9]
Statistical Analysis 9: Comparison: 0.75 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison for HbA1c less than or equal to 6.5%; Odds Ratio (OR) = 2.4, 95% CI 2-sided [1.6 to 3.5]
Statistical Analysis 10: Comparison: Exenatide vs Placebo; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison for HbA1c less than or equal to 6.5%; Odds Ratio (OR) = 2.7, 95% CI 2-sided [1.6 to 4.6]

10. Secondary Outcome: Percentage of Participants Attaining Glycosylated Hemoglobin (HbA1c) Less Than 7% and Less Than or Equal to 6.5% at 52 Weeks
Description: as for outcome 9
Time Frame: Baseline, 52 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide
Number analyzed (Participants) | 271 | 269 | 266
percentage of participants
  HbA1c Less Than 7.0% | 70.8 | 59.1 | 49.2
  HbA1c Less Than or Equal to 6.5% | 57.2 | 48.3 | 34.6
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison for HbA1c less than 7.0%; Odds Ratio (OR) = 3.7, 95% CI 2-sided [2.4 to 5.6]
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p = 0.008, Regression, Logistic — Treatment comparison for HbA1c less than 7.0%; Odds Ratio (OR) = 1.7, 95% CI 2-sided [1.1 to 2.5]
Statistical Analysis 3: Comparison: 1.5 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison for HbA1c less than or equal to 6.5%; Odds Ratio (OR) = 3.5, 95% CI 2-sided [2.3 to 5.1]
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison for HbA1c less than or equal to 6.5%; Odds Ratio (OR) = 2.1, 95% CI 2-sided [1.4 to 3.1]

11. Secondary Outcome: Change From Baseline to 26 Weeks in Updated Homeostasis Model Assessment of Beta-cell Function (HOMA2-%B) and Updated Homeostasis Model Assessment of Insulin Sensitivity (HOMA2-%S)
Description: The homeostatic model assessment (HOMA) quantifies insulin resistance and beta-cell function. HOMA2-B is a computer model that uses fasting plasma insulin and glucose concentrations to estimate steady-state beta cell function (%B) as a percentage of a normal reference population (normal young adults). HOMA2-S is a computer model that uses fasting plasma insulin and glucose concentrations to estimate insulin sensitivity (%S) as percentages of a normal reference population (normal young adults). The normal reference populations were set at 100%. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265, Exenatide, or Placebo with evaluable HOMA2-%B or HOMA2-%S data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: percentage of HOMA2
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 238 | 218 | 223 | 98
percentage of HOMA2
  HOMA2-%B | 36.14 (2.60) | 23.61 (2.67) | 15.02 (2.62) | 0.93 (3.66)
  HOMA2-%S | -3.14 (2.91) | 1.16 (2.97) | -1.59 (2.92) | 2.56 (4.07)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of HOMA2-B; LS Mean Difference = 35.21, 95% CI 2-sided [27.26 to 43.16]
Statistical Analysis 2: Comparison: 1.5 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of HOMA2-B; LS Mean Difference = 21.12, 95% CI 2-sided [14.97 to 27.28]
Statistical Analysis 3: Comparison: 0.75 mg LY2189265 vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of HOMA2-B; LS Mean Difference = 22.68, 95% CI 2-sided [14.63 to 30.72]
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis — Treatment comparison of HOMA2-B; LS Mean Difference = 8.59, 95% CI 2-sided [2.31 to 14.87]
Statistical Analysis 5: Comparison: Exenatide vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of HOMA2-B; LS Mean Difference = 14.09, 95% CI 2-sided [6.06 to 22.11]
Statistical Analysis 6: Comparison: 1.5 mg LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.207, Mixed Models Analysis — Treatment comparison of HOMA2-S; LS Mean Difference = -5.70, 95% CI 2-sided [-14.56 to 3.17]
Statistical Analysis 7: Comparison: 1.5 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p = 0.659, Mixed Models Analysis — Treatment comparison of HOMA2-S; LS Mean Difference = -1.54, 95% CI 2-sided [-8.41 to 5.32]
Statistical Analysis 8: Comparison: 0.75 mg LY2189265 vs Placebo; Test type: Superiority or Other; p = 0.759, Mixed Models Analysis — Treatment comparison of HOMA2-S; LS Mean Difference = -1.40, 95% CI 2-sided [-10.37 to 7.56]
Statistical Analysis 9: Comparison: 0.75 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p = 0.441, Mixed Models Analysis — Treatment comparison of HOMA2-S; LS Mean Difference = 2.75, 95% CI 2-sided [-4.25 to 9.76]
Statistical Analysis 10: Comparison: Exenatide vs Placebo; Test type: Superiority or Other; p = 0.362, Mixed Models Analysis — Treatment comparison of HOMA2-S; LS Mean Difference = -4.15, 95% CI 2-sided [-13.10 to 4.79]

12. Secondary Outcome: Change From Baseline to 52 Weeks in Updated Homeostasis Model Assessment of Beta-cell Function (HOMA2-%B) and Updated Homeostasis Model Assessment of Insulin Sensitivity (HOMA2-%S)
Description: as for outcome 11
Time Frame: Baseline, 52 weeks
Population: Participants who were randomized at baseline to LY2189265 or Exenatide and received at least 1 dose of study drug with evaluable HOMA2-%B or HOMA2-%S data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: percentage of HOMA2
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide
Number analyzed (Participants) | 219 | 202 | 187
percentage of HOMA2
  HOMA2-%B | 35.21 (2.63) | 25.69 (2.70) | 13.57 (2.75)
  HOMA2-%S | -7.48 (2.93) | -5.49 (3.01) | -3.75 (3.07)
Statistical Analysis 1: Comparison: 1.5 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of HOMA2-B; LS Mean Difference = 21.64, 95% CI 2-sided [15.20 to 28.08]
Statistical Analysis 2: Comparison: 0.75 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Treatment comparison of HOMA2-B; LS Mean Difference = 12.12, 95% CI 2-sided [5.56 to 18.68]
Statistical Analysis 3: Comparison: 1.5 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p = 0.307, Mixed Models Analysis — Treatment comparison of HOMA2-S; LS Mean Difference = -3.73, 95% CI 2-sided [-10.90 to 3.43]
Statistical Analysis 4: Comparison: 0.75 mg LY2189265 vs Exenatide; Test type: Superiority or Other; p = 0.638, Mixed Models Analysis — Treatment comparison of HOMA2-S; LS Mean Difference = -1.75, 95% CI 2-sided [-9.05 to 5.55]

13. Secondary Outcome: Change From Baseline to 26 Weeks in the EuroQol 5
Description: The European Quality of Life - 5 dimensions (EQ-5D) questionnaire is a generic, multidimensional, health-related, quality-of-life instrument. It consists of 2 parts: the first part assesses 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) that have 3 possible levels of response (no problem, some problem, or extreme problem). These dimensions are converted into a weighted health-state Index Score. The EQ-5D United Kingdom (UK) score ranges from -0.59 to 1.0, where a score of 1.0 indicates perfect health and negative values are valued as worse than dead. The second part of the questionnaire consists of a visual analog scale (VAS) on which the participants rated their perceived health state on that day from 0 (worst imaginable health state) to 100 (best imaginable health). Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) and adjusted by treatment, country, and baseline.
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265, Exenatide, or Placebo with evaluable EQ-5D data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 279 | 280 | 276 | 141
units on a scale
  VAS Health State Score (n=270, 267, 264, 119) | 4.50 (0.85) | 2.41 (0.85) | 3.94 (0.85) | 0.71 (1.15)
  EQ-5D UK (n=270, 266, 264, 119) | 0.01 (0.01) | 0.01 (0.01) | 0.00 (0.01) | -0.00 (0.02)

14. Secondary Outcome: Change From Baseline to 52 Weeks in the EuroQol 5
Description: as for outcome 13
Time Frame: Baseline, 52 weeks
Population: Participants who were randomized at baseline to LY2189265 or Exenatide and received at least 1 dose of study drug with evaluable EQ-5D data. Only pre-rescue measurements were used. LOCF was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide
Number analyzed (Participants) | 279 | 280 | 276
units on a scale
  VAS Health State Score (n=270, 267, 264) | 5.15 (0.89) | 3.52 (0.89) | 3.51 (0.89)
  EQ-5D UK (n=270, 266, 264) | 0.02 (0.01) | 0.01 (0.01) | -0.00 (0.01)

15. Secondary Outcome: Change From Baseline to 26 Weeks in the Diabetes Treatment Satisfaction Questionnaire Status (DTSQs) Version
Description: The Diabetes Treatment Satisfaction Questionnaire status version (DTSQs) is used to assess participant treatment satisfaction at each study visit. The questionnaire consists of 8 items, 6 of which (1, and 4 through 8) assess treatment satisfaction. Each item is rated on a 7-point Likert scale. Scores from the 6 treatment satisfaction items are summed to a Total Treatment Satisfaction Score, which ranges from 0 (very dissatisfied) to 36 (very satisfied). The DTSQ change version (DTSQc) was not collected at 26 weeks. Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) with country and treatment as fixed effects and baseline score as a covariate.
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265, Exenatide, or Placebo with evaluable DTSQs data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) used to impute missing postbaseline values. If there were no data after randomization, endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 270 | 268 | 266 | 119
units on a scale | 2.40 (0.34) | 2.56 (0.33) | 0.85 (0.33) | 0.49 (0.45)

16. Secondary Outcome: Change From Baseline to 52 Weeks in the Diabetes Treatment Satisfaction Questionnaire Status (DTSQs) and Change (DTSQc) Versions
Description: The Diabetes Treatment Satisfaction Questionnaire status (DTSQs) and change (DTSQc) versions are used to assess participant treatment satisfaction at each study visit and relative change in satisfaction from baseline, respectively. Both questionnaires consist of 8 items, 6 of which (1, and 4 through 8) assess treatment satisfaction. Each item is rated on a 7-point Likert scale. The change version has the same 8 items as the status version with a small alteration of the wording of Item 7. Scores from the 6 treatment satisfaction items are summed to a Total Treatment Satisfaction Score, which ranges from 0 (very dissatisfied) to 36 (very satisfied) for the DTSQs and from -18 (much less satisfied) to +18 (much more satisfied) for the DTSQc. Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) with country and treatment as fixed effects and baseline score as a covariate.
Time Frame: Baseline, 52 weeks
Population: Participants who were randomized at baseline to LY2189265 or Exenatide and received at least 1 dose of study drug with evaluable DTSQs or DTSQc data. Only pre-rescue measurements were used. LOCF was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide
Number analyzed (Participants) | 279 | 280 | 276
units on a scale
  DTSQs Treatment Satisfaction (n=270, 268, 266) | 2.05 (0.36) | 2.11 (0.36) | 0.69 (0.36)
  DTSQc Treatment Satisfaction (n=249, 237, 226) | 15.36 (0.40) | 15.46 (0.41) | 14.01 (0.41)

17. Secondary Outcome: Change From Baseline to 26 Weeks in the Impact of Weight on Activities of Daily Living
Description: The Impact of Weight on Activities of Daily Living (renamed the Ability to Perform Physical Activities of Daily Living [APPADL]) questionnaire contains 7 items that assess how difficult it is for participants to engage in certain activities considered to be integral to normal daily life, such as walking, standing and climbing stairs. Items are scored on a 5-point numeric rating scale where 5 = "not at all difficult" and 1 = "unable to do". The individual scores from all 7 items are summed and a single total score is calculated and may range between 7 and 35. A higher score indicates better ability to perform activities of daily living. Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) with country and treatment as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265, Exenatide, or Placebo with evaluable APPADL data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 270 | 267 | 266 | 119
units on a scale | 0.18 (0.27) | 0.12 (0.27) | 0.47 (0.27) | 0.03 (0.36)

18. Secondary Outcome: Change From Baseline to 52 Weeks in the Impact of Weight on Activities of Daily Living
Description: as for outcome 17
Time Frame: Baseline, 52 weeks
Population: Participants who were randomized at baseline to LY2189265 or Exenatide and received at least 1 dose of study drug with evaluable APPADL data. Only pre-rescue measurements were used. LOCF was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide
Number analyzed (Participants) | 270 | 267 | 266
units on a scale | 0.18 (0.29) | -0.18 (0.29) | 0.35 (0.29)

19. Secondary Outcome: Change From Baseline to 26 Weeks on the Impact of Weight on Self-Perception
Description: The Impact of Weight on Self-Perception (IW-SP) questionnaire contains 3 items that assess how often the participants' body weight affects how happy they are with their appearance and how often they feel self-conscious when out in public. Items are scored on a 5-point numeric rating scale where 5 = never and 1 = always. A single total score is calculated by summing the scores for all 3 items. Total score ranges between 3 and 15, where a higher score is indicative of better self-perception. Least Squares (LS) means of change from baseline were calculated using analysis of covariance (ANCOVA) with country and treatment as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265, Exenatide, or Placebo with evaluable IW-SP data. Only pre-rescue measurements were used. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 270 | 267 | 266 | 119
units on a scale | 0.56 (0.15) | 0.47 (0.15) | 0.46 (0.15) | 0.45 (0.20)

20. Secondary Outcome: Change From Baseline to 52 Weeks on the Impact of Weight on Self-Perception
Description: as for outcome 19
Time Frame: Baseline, 52 weeks
Population: Participants who were randomized at baseline to LY2189265 or Exenatide and received at least 1 dose of study drug with evaluable IW-SP data. Only pre-rescue measurements were used. LOCF was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide
Number analyzed (Participants) | 270 | 267 | 266
units on a scale | 0.50 (0.15) | 0.47 (0.15) | 0.64 (0.15)

21. Secondary Outcome: Number of Participants With Adjudicated Cardiovascular Events at 52 Weeks
Description: Information on cardiovascular (CV) risk factors was collected at baseline. Data on any new CV event was prospectively collected using a CV event electronic case report form. At prespecified visits, participants were asked about any new CV event since the previous inquiry. Deaths and nonfatal cardiovascular adverse events (AEs) were adjudicated by an external committee of physicians with cardiology expertise. Nonfatal cardiovascular AEs to be adjudicated included myocardial infarction, hospitalization for unstable angina, hospitalization for heart failure, coronary interventions, and cerebrovascular events, including cerebrovascular accident (stroke) and transient ischemic attack. The number of participants with CV events confirmed by adjudication is summarized cumulatively at 52 weeks. Serious and all other non-serious adverse events regardless of causality are summarized in the Reported Adverse Events module.
Time Frame: Baseline through 52 weeks
Population: Participants who were randomized at baseline to LY2189265 or Exenatide and received at least 1 dose of study drug. The number of participants with adjudicated CV events was not collected at 26 weeks.
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide
Number analyzed (Participants) | 279 | 280 | 276
participants
  Any CV Event | 3 | 2 | 2
  Any Fatal Event | 1 | 0 | 0
  Any Non-fatal CV Event | 3 | 2 | 2

22. Secondary Outcome: Change From Baseline to 26 Weeks on Electrocardiogram Parameters, Fridericia Corrected QT (QTcF) Interval and PR Interval
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave and was calculated from electrocardiogram (ECG) data using Fridericia's formula: QTc = QT/RR^0.33. Corrected QT (QTc) is the QT interval corrected for heart rate and RR, which is the interval between two R waves. PR is the interval between the P wave and the QRS complex. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265, Exenatide, or Placebo with evaluable ECG QTcF Interval or PR interval data.
Measure: Least Squares Mean (Standard Error); unit: milliseconds (msec)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 279 | 280 | 276 | 141
milliseconds (msec)
  QTcF Interval (n=253, 260, 250, 120) | -1.11 (1.00) | 0.91 (0.99) | 1.21 (1.00) | 1.32 (1.33)
  PR Interval (n=252, 259, 246, 116) | 2.35 (0.89) | 0.93 (0.88) | 1.01 (0.89) | -1.83 (1.20)

23. Secondary Outcome: Change From Baseline to 52 Weeks on Electrocardiogram Parameters, Fridericia Corrected QT (QTcF) Interval and PR Interval
Description: as for outcome 22
Time Frame: Baseline, 52 weeks
Population: Participants who were randomized at baseline to LY2189265 or Exenatide and received at least 1 dose of study drug with evaluable ECG QTcF Interval or PR Interval data.
Measure: Least Squares Mean (Standard Error); unit: milliseconds (msec)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide
Number analyzed (Participants) | 279 | 280 | 276
milliseconds (msec)
  QTcF Interval (n=239, 243, 226) | 1.28 (1.07) | 2.30 (1.07) | 2.52 (1.10)
  PR Interval (n=237, 243, 220) | 2.57 (0.96) | 0.69 (0.96) | -0.82 (0.99)

24. Secondary Outcome: Change in Baseline to 26 Weeks on Pulse Rate
Description: Seated pulse rate was measured. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265, Exenatide, or Placebo with evaluable seated pulse rate data.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 263 | 266 | 259 | 127
beats per minute (bpm) | 2.80 (0.52) | 2.80 (0.51) | 1.18 (0.52) | 0.61 (0.70)

25. Secondary Outcome: Change in Baseline to 52 Weeks on Pulse Rate
Description: as for outcome 24
Time Frame: Baseline, 52 weeks
Population: Participants who were randomized at baseline to LY2189265 or Exenatide and received at least 1 dose of study drug with evaluable seated pulse rate data.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide
Number analyzed (Participants) | 248 | 256 | 238
beats per minute (bpm) | 1.68 (0.56) | 1.56 (0.55) | 1.15 (0.56)

26. Secondary Outcome: Change From Baseline to 26 Weeks on Blood Pressure
Description: Seated systolic blood pressure (SBP) and seated diastolic blood pressure (DBP) were measured. Least Squares (LS) means of change from baseline were calculated using a mixed-effects model for repeated measures (MMRM) with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized and received at least one dose of LY2189265, Exenatide, or Placebo with evaluable blood pressure data.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 279 | 280 | 276 | 141
millimeters of mercury (mmHg)
  Seated SBP (n=263, 266, 259, 127) | 0.11 (0.83) | -0.36 (0.82) | 0.06 (0.83) | 3.40 (1.13)
  Seated DBP (n=263, 266, 259, 127) | 0.76 (0.55) | 0.56 (0.54) | -0.11 (0.55) | 1.25 (0.75)

27. Secondary Outcome: Change From Baseline to 52 Weeks on Blood Pressure
Description: as for outcome 26
Time Frame: Baseline, 52 weeks
Population: Participants who were randomized at baseline to LY2189265 or Exenatide and received at least 1 dose of study drug with evaluable blood pressure data.
Measure: Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide
Number analyzed (Participants) | 279 | 280 | 276
millimeters of mercury (mmHg)
  Seated SBP (n=248, 256, 238) | 0.83 (0.87) | 1.62 (0.85) | 0.02 (0.88)
  Seated DBP (n=248, 256, 238) | 0.89 (0.57) | 0.76 (0.57) | 0.02 (0.58)

28. Secondary Outcome: Number of Participants With Adjudicated Pancreatitis at 26 Weeks
Description: The number of participants with pancreatitis confirmed by adjudication is summarized cumulatively at 26 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265, Exenatide, or Placebo.
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 279 | 280 | 276 | 141
participants | 0 | 0 | 0 | 0

29. Secondary Outcome: Number of Participants With Adjudicated Pancreatitis at 52 Weeks
Description: The number of participants with pancreatitis confirmed by adjudication is summarized cumulatively at 52 weeks, with the exception of the Placebo/1.5 mg LY2189265 and Placebo/0.75 mg LY2189265 treatment groups, which include only participants with confirmed pancreatitis during treatment with LY2189265 (26 weeks through 52 weeks). A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 52 weeks
Population: Participants who were randomized at baseline to LY2189265, Exenatide, or Placebo and received at least 1 dose of study drug.
Measure: Number; unit: participants
Groups:
- Placebo/1.5 mg LY2189265: Placebo: subcutaneous (SC), once weekly for 26 weeks
  LY2189265 (Dulaglutide): 1.5 milligrams (mg), SC, once weekly from week 26 through week 52
  Metformin: at least 1500 milligrams per day (mg/day), oral, for 52 weeks
  Pioglitazone: at least 30 mg/day, oral, for 52 weeks
- Placebo/0.75 mg LY2189265: Placebo: subcutaneous (SC), once weekly for 26 weeks
  LY2189265 (Dulaglutide): 0.75 milligrams (mg), SC, once weekly from week 26 through week 52
  Metformin: at least 1500 milligrams per day (mg/day), oral, for 52 weeks
  Pioglitazone: at least 30 mg/day, oral, for 52 weeks
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo/1.5 mg LY2189265 | Placebo/0.75 mg LY2189265
Number analyzed (Participants) | 279 | 280 | 276 | 62 | 62
participants | 1 | 0 | 0 | 0 | 0

30. Secondary Outcome: Change From Baseline to 26 Weeks on Pancreatic Enzymes
Description: Amylase (total and pancreas-derived) and lipase concentrations were measured.
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265, Exenatide, or Placebo with evaluable pancreatic enzyme data. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Median (Inter-Quartile Range); unit: units per liter
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 279 | 280 | 276 | 141
units per liter
  Amylase, Total (n=253, 253, 254, 127) | 12.50 (26.55) [-3.57 to 28.85] | 3.28 (24.24) [-9.88 to 20.00] | 5.56 (26.61) [-9.52 to 18.46] | -3.33 (27.51) [-15.79 to 11.36]
  Amylase, Pancreas-derived (n=237, 247, 246, 122) | 14.81 [0.00 to 35.00] | 10.34 [-5.88 to 26.67] | 5.56 [-7.14 to 21.05] | -3.77 [-13.33 to 13.64]
  Lipase (n=198, 203, 222, 114) | 10.34 [-7.50 to 29.41] | 0.00 [-15.91 to 23.08] | 3.94 [-10.26 to 23.08] | -9.53 [-23.33 to 6.67]

31. Secondary Outcome: Change From Baseline to 52 Weeks on Pancreatic Enzymes
Description: Amylase (total and pancreas-derived) and lipase concentrations were measured.
Time Frame: Baseline, 52 weeks
Population: Participants who were randomized at baseline to LY2189265 or Exenatide and received at least 1 dose of study drug with evaluable pancreatic enzyme data. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Median (Inter-Quartile Range); unit: units per liter
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide
Number analyzed (Participants) | 279 | 280 | 276
units per liter
  Amylase, Total (n=255, 263, 261) | 9.21 [-4.95 to 23.19] | 2.78 [-11.67 to 17.50] | 2.38 [-11.86 to 15.22]
  Amylase, Pancreas-derived (n=236, 253, 246) | 16.67 [0.00 to 35.60] | 7.69 [-8.70 to 28.00] | 7.85 [-8.82 to 26.67]
  Lipase (n=201, 205, 221) | 5.45 [-7.69 to 26.92] | 0.00 [-18.18 to 15.63] | 3.57 [-13.95 to 22.58]

32. Secondary Outcome: Change From Baseline to 26 Weeks on Serum Calcitonin
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265, Exenatide, or Placebo with evaluable serum calcitonin data. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 275 | 277 | 272 | 139
picograms per milliliter (pg/mL) | 0.20 (1.20) | 0.22 (1.91) | 0.05 (1.48) | 0.05 (0.89)

33. Secondary Outcome: Change From Baseline to 52 Weeks on Serum Calcitonin
Time Frame: Baseline, 52 weeks
Population: Participants who were randomized at baseline to LY2189265 or Exenatide and received at least 1 dose of study drug with evaluable serum calcitonin data. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide
Number analyzed (Participants) | 275 | 277 | 272
picograms per milliliter (pg/mL) | 0.21 (1.29) | 0.05 (1.79) | 0.10 (1.67)

34. Secondary Outcome: Number of Self-reported Hypoglycemic Events at 26 Weeks
Description: Hypoglycemic events (HE) were classified as severe (defined as episodes requiring the assistance of another person to actively administer resuscitative actions), documented symptomatic (defined as any time a participant feels that he/she is experiencing symptoms and/or signs associated with hypoglycemia, and has a plasma glucose level of less than or equal to 3.9 millimoles/liter [mmol/L]), asymptomatic (defined as events not accompanied by typical symptoms of hypoglycemia but with a measured plasma glucose of less than or equal to 3.9 mmol/L), nocturnal (defined as any hypoglycemic event that occurred between bedtime and waking), or probable symptomatic (defined as events during which symptoms of hypoglycemia were not accompanied by a plasma glucose determination). The number of self-reported hypoglycemic events is summarized cumulatively at 26 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265, Exenatide, or Placebo.
Measure: Number; unit: events
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 279 | 280 | 276 | 141
events
  Severe HE | 0 | 0 | 1 | 0
  Documented Symptomatic HE | 31 | 25 | 146 | 4
  Asymptomatic HE | 26 | 95 | 51 | 5
  Nocturnal HE | 9 | 15 | 31 | 6
  Probable Symptomatic HE | 5 | 16 | 3 | 3

35. Secondary Outcome: Number of Self-reported Hypoglycemic Events at 52 Weeks
Description: Hypoglycemic events (HE) were classified as severe (defined as episodes requiring the assistance of another person to actively administer resuscitative actions), documented symptomatic (defined as any time a participant feels that he/she is experiencing symptoms and/or signs associated with hypoglycemia, and has a plasma glucose level of less than or equal to 3.9 millimoles/liter [mmol/L]), asymptomatic (defined as events not accompanied by typical symptoms of hypoglycemia but with a measured plasma glucose of less than or equal to 3.9 mmol/L), nocturnal (defined as any hypoglycemic event that occurred between bedtime and waking), or probable symptomatic (defined as events during which symptoms of hypoglycemia were not accompanied by a plasma glucose determination). The number of self-reported hypoglycemic events is summarized cumulatively at 52 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 52 weeks
Population: Participants who were randomized at baseline to LY2189265 or Exenatide and received at least 1 dose of study drug.
Measure: Number; unit: events
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide
Number analyzed (Participants) | 279 | 280 | 276
events
  Severe HE | 0 | 0 | 2
  Documented Symptomatic HE | 53 | 39 | 205
  Asymptomatic HE | 47 | 157 | 98
  Nocturnal HE | 20 | 29 | 57
  Probable Symptomatic HE | 8 | 22 | 4

36. Secondary Outcome: Rate of Self-reported Hypoglycemic Events at 26 Weeks
Description: Hypoglycemic events (HE) were classified as severe (defined as episodes requiring the assistance of another person to actively administer resuscitative actions), documented symptomatic (defined as any time a participant feels that he/she is experiencing symptoms and/or signs associated with hypoglycemia, and has a plasma glucose level of equal to or less than 3.9 millimoles/liter [mmol/L]), asymptomatic (defined as events not accompanied by typical symptoms of hypoglycemia but with a measured plasma glucose of equal to or less than 3.9 mmol/L), nocturnal (defined as any hypoglycemic event that occurred between bedtime and waking), or probable symptomatic (defined as events during which symptoms of hypoglycemia were not accompanied by a plasma glucose determination). The 1-year adjusted rate of hypoglycemic events is summarized cumulatively at 26 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 weeks
Population: Participants who were randomized and received at least one dose of LY2189265, Exenatide, or Placebo. Only pre-rescue measurements were used.
Measure: Mean (Standard Deviation); unit: events per participant per year
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 279 | 280 | 276 | 141
events per participant per year
  Severe HE | 0.00 (0.00) | 0.00 (0.00) | 0.01 (0.12) | 0.00 (0.00)
  Documented symptomatic HE | 0.22 (1.94) | 0.18 (0.97) | 1.07 (4.90) | 0.06 (0.48)
  Asymptomatic HE | 0.19 (1.13) | 0.69 (4.74) | 0.38 (1.74) | 0.27 (2.44)
  Nocturnal HE | 0.06 (0.60) | 0.19 (1.74) | 0.23 (1.16) | 0.27 (2.51)
  Probable symptomatic HE | 0.04 (0.37) | 0.24 (2.44) | 0.02 (0.21) | 0.04 (0.51)

37. Secondary Outcome: Rate of Self-reported Hypoglycemic Events at 52 Weeks
Description: Hypoglycemic events (HE) were classified as severe (defined as episodes requiring the assistance of another person to actively administer resuscitative actions), documented symptomatic (defined as any time a participant feels that he/she is experiencing symptoms and/or signs associated with hypoglycemia, and has a plasma glucose level of equal to or less than millimoles/liter [mmol/L]), asymptomatic (defined as events not accompanied by typical symptoms of hypoglycemia but with a measured plasma glucose of equal to or less than 3.9 mmol/L), nocturnal (defined as any hypoglycemic event that occurred between bedtime and waking), or probable symptomatic (defined as events during which symptoms of hypoglycemia were not accompanied by a plasma glucose determination). The 1-year adjusted rate of hypoglycemic events is summarized cumulatively at 52 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 52 weeks
Population: Participants who were randomized at baseline to LY2189265 or Exenatide and received at least 1 dose of study drug. Only pre-rescue measurements were used.
Measure: Mean (Standard Deviation); unit: events per participant per year
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide
Number analyzed (Participants) | 279 | 280 | 276
events per participant per year
  Severe HE | 0.00 (0.00) | 0.00 (0.00) | 0.01 (0.09)
  Documented symptomatic HE | 0.19 (1.23) | 0.14 (0.78) | 0.76 (3.18)
  Asymptomatic HE | 0.17 (1.05) | 0.56 (3.57) | 0.37 (1.81)
  Nocturnal HE | 0.07 (0.63) | 0.19 (1.72) | 0.21 (1.06)
  Probable symptomatic HE | 0.03 (0.26) | 0.21 (2.38) | 0.02 (0.16)

38. Secondary Outcome: Number of Participants Requiring Rescue Therapy Due to Hyperglycemia at 26 Weeks
Description: Rescue therapy was defined as any additional therapeutic intervention in participants who developed persistent, severe hyperglycemia despite full compliance with the assigned therapeutic regimen, or initiation of an alternative antihyperglycemic medication following study drug discontinuation. Participants who had no rescue therapy within specified study period were considered as censored observations at the last available contact date up to specified study period. Time to start first new glucose-lowering intervention due to hyperglycemia ("rescue therapy") was analyzed between the groups using the semi-parametric proportional hazard regression model with treatment group and country as fixed effects and baseline glycosylated hemoglobin (HbA1c) as a covariate.
Time Frame: Baseline through 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265, Exenatide, or Placebo.
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 279 | 280 | 276 | 141
participants | 4 | 14 | 13 | 22

39. Secondary Outcome: Number of Participants Requiring Rescue Therapy Due to Hyperglycemia at 52 Weeks
Description: as for outcome 38
Time Frame: Baseline through 52 weeks
Population: Participants who were randomized at baseline to LY2189265 or Exenatide and received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide
Number analyzed (Participants) | 279 | 280 | 276
participants | 10 | 27 | 31

40. Secondary Outcome: Number of Participants With LY2189265 Antibodies at 26 Weeks
Description: LY2189265 (Dulaglutide) anti-drug antibodies (ADA) were assessed. The number of participants with initial postbaseline detection of treatment emergent (defined as a 4-fold increase in the ADA titer from baseline) LY2189265 ADA were summarized.
Time Frame: Baseline through 26 weeks
Population: Participants who were randomized and received at least one dose of LY2189265, Exenatide, or Placebo with evaluable LY2189265 ADA data. In the clinically evaluated dose range of LY2189265, no dose effect on the magnitude of the anti-LY2189265 immune response was observed. Therefore, results were combined for the 0.75 mg and 1.5 mg LY2189265 groups.
Measure: Number; unit: participants
Groups:
- 0.75 mg LY2189265 or 1.5 mg LY2189265: LY2189265 (Dulaglutide): 0.75 or 1.5 milligrams (mg), subcutaneous (SC), once weekly for 52 weeks
  Metformin: at least 1500 milligrams per day (mg/day), oral, for 52 weeks
  Pioglitazone: at least 30 mg/day, oral, for 52 weeks
Arm/Group | 0.75 mg LY2189265 or 1.5 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 559 | 276 | 141
participants | 6 | 12 | 2

41. Secondary Outcome: Number of Participants With LY2189265 Antibodies at 52 Weeks and 4 Weeks After Last Dose of Study Drug
Description: as for outcome 40
Time Frame: 26 weeks through 52 weeks and 53 weeks through 4 weeks after last dose
Population: as for outcome 40
Measure: Number; unit: participants
Groups:
- Placebo/0.75 mg LY2189265 or 1.5 mg LY2189265: Placebo: subcutaneous (SC), once weekly for 26 weeks
  LY2189265 (Dulaglutide): 0.75 or 1.5 milligrams (mg), SC, once weekly from week 26 through week 52
  Metformin: at least 1500 milligrams per day (mg/day), oral, for 52 weeks
  Pioglitazone: at least 30 mg/day, oral, for 52 weeks
Arm/Group | 0.75 mg LY2189265 or 1.5 mg LY2189265 | Exenatide | Placebo/0.75 mg LY2189265 or 1.5 mg LY2189265
Number analyzed (Participants) | 552 | 270 | 123
participants
  52 weeks | 3 | 2 | 2
  4 weeks after last study dose | 1 | 0 | 1

42. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events at 26 Weeks
Description: A treatment-emergent adverse event (TEAE) was defined as an event that first occurs or worsens (increases in severity) after baseline regardless of causality or severity. The number of participants with one or more TEAE is summarized cumulatively at 26 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265, Exenatide, or Placebo.
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 279 | 280 | 276 | 141
participants | 215 | 199 | 198 | 104

43. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events at 52 Weeks
Description: A treatment-emergent adverse event (TEAE) was defined as an event that first occurs or worsens (increases in severity) after baseline regardless of causality or severity. The number of participants with one or more TEAE is summarized cumulatively at 52 weeks, with the exception of the Placebo/1.5 mg LY2189265 and Placebo/0.75 mg LY2189265 treatment groups, which include only TEAEs that occurred during treatment with LY2189265 (26 weeks through 52 weeks). A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 52 weeks
Population: as for outcome 29
Measure: Number; unit: participants
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo/1.5 mg LY2189265 | Placebo/0.75 mg LY2189265
Number analyzed (Participants) | 279 | 280 | 276 | 62 | 62
participants | 226 | 220 | 221 | 47 | 41

44. Secondary Outcome: Change From Baseline to 26 Weeks in Hematological and Biochemical Lab Values
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265, Exenatide, or Placebo.
Measure: Least Squares Mean (Standard Error)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 279 | 280 | 276 | 141
Value | NA (NA) — No clinically relevant changes from baseline to 26 weeks in hematological and biochemical laboratory values were noted, with the exception of pancreatic enzymes and calcitonin measures, which are reported in separate outcome measures. | NA (NA) — No clinically relevant changes from baseline to 26 weeks in hematological and biochemical laboratory values were noted, with the exception of pancreatic enzymes and calcitonin measures, which are reported in separate outcome measures. | NA (NA) — No clinically relevant changes from baseline to 26 weeks in hematological and biochemical laboratory values were noted, with the exception of pancreatic enzymes and calcitonin measures, which are reported in separate outcome measures. | NA (NA) — No clinically relevant changes from baseline to 26 weeks in hematological and biochemical laboratory values were noted, with the exception of pancreatic enzymes and calcitonin measures, which are reported in separate outcome measures.

45. Secondary Outcome: Change From Baseline to 52 Weeks in Hematological and Biochemical Lab Values
Time Frame: Baseline, 52 weeks
Population: Participants who were randomized at baseline to LY2189265 or Exenatide and received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide
Number analyzed (Participants) | 279 | 280 | 276
Value | NA (NA) — No clinically relevant changes from baseline to 26 weeks in hematological and biochemical laboratory values were noted, with the exception of pancreatic enzymes and calcitonin measures, which are reported in separate outcome measures. | NA (NA) — No clinically relevant changes from baseline to 26 weeks in hematological and biochemical laboratory values were noted, with the exception of pancreatic enzymes and calcitonin measures, which are reported in separate outcome measures. | NA (NA) — No clinically relevant changes from baseline to 26 weeks in hematological and biochemical laboratory values were noted, with the exception of pancreatic enzymes and calcitonin measures, which are reported in separate outcome measures.

46. Secondary Outcome: Change From Baseline to 26 Weeks in N Terminal Pro Brain Natriuretic Peptide (NT-proBNP)
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265, Exenatide, or Placebo with evaluable NT-proBNP data. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Median (Inter-Quartile Range); unit: picograms per milliliter (pg/mL)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265 | Exenatide | Placebo
Number analyzed (Participants) | 255 | 254 | 246 | 119
picograms per milliliter (pg/mL) | -6.77 (91.13) [-30.45 to 15.22] | -2.96 (189.94) [-22.83 to 19.45] | -3.38 (208.92) [-31.29 to 18.61] | -0.85 (133.04) [-25.37 to 17.76]

47. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve (AUC) for LY2189265
Description: Evaluable pharmacokinetic concentrations from the 4-week, 13-week, 26-week, and 52-week timepoints were combined and utilized in a population approach to determine the population mean estimate and standard deviation at steady-state.
Time Frame: 4 weeks, 13 weeks, 26 weeks, and 52 weeks
Population: Participants who were randomized at baseline to LY2189265 and received at least 1 dose of study drug with evaluable AUC data.
Measure: Mean (Standard Deviation); unit: nanogram hours per milliliter (ng*hr/mL)
Arm/Group | 1.5 mg LY2189265 | 0.75 mg LY2189265
Number analyzed (Participants) | 325 | 321
nanogram hours per milliliter (ng*hr/mL) | 12383 (5433) | 6627 (2487)

ADVERSE EVENTS:
Groups:
- 0.75 mg LY2189265 (Baseline Through 26 Weeks); 0.75 mg LY2189265 (Baseline Through 56 Weeks): LY2189265 (Dulaglutide): 0.75 milligrams (mg), subcutaneous (SC), once weekly for 52 weeks
  Metformin: at least 1500 milligrams per day (mg/day), oral, for 52 weeks
  Pioglitazone: at least 30 mg/day, oral, for 52 weeks
- 1.5 mg LY2189265 (Baseline Through 26 Weeks); 1.5 mg LY2189265 (Baseline Through 56 Weeks): LY2189265 (Dulaglutide): 1.5 milligrams (mg), subcutaneous (SC), once weekly for 52 weeks
  Metformin: at least 1500 milligrams per day (mg/day), oral, for 52 weeks
  Pioglitazone: at least 30 mg/day, oral, for 52 weeks
- Exenatide (Baseline Through 26 Weeks); Exenatide (Baseline Through 56 Weeks): Exenatide: 5 micrograms (mcg), subcutaneous (SC), twice daily for 4 weeks, followed by 10 mcg, SC, twice daily for 48 weeks
  Metformin: at least 1500 milligrams per day (mg/day), oral, for 52 weeks
  Pioglitazone: at least 30 mg/day, oral, for 52 weeks
- Placebo (Baseline Through 26 Weeks): Placebo: subcutaneous (SC), once weekly for 26 weeks
  LY2189265 (Dulaglutide): After 26 weeks, participants were randomized to receive either 0.75 milligrams (mg) or 1.5 mg, SC, once weekly for an additional 26 weeks (from week 26 through week 52)
  Metformin: at least 1500 milligrams per day (mg/day), oral, for 52 weeks
  Pioglitazone: at least 30 mg/day, oral, for 52 weeks
- Placebo/0.75 mg LY2189265 (26 Weeks Through 56 Weeks): Placebo: subcutaneous (SC), once weekly for 26 weeks
  LY2189265 (Dulaglutide): 0.75 milligrams (mg), SC, once weekly from week 26 through week 52
  Metformin: at least 1500 milligrams per day (mg/day), oral, for 52 weeks
  Pioglitazone: at least 30 mg/day, oral, for 52 weeks
  All events were treatment emergent during the LY2189265 treatment period.
- Placebo/1.5 mg LY2189265 (26 Weeks Through 56 Weeks): Placebo: subcutaneous (SC), once weekly for 26 weeks
  LY2189265 (Dulaglutide): 1.5 milligrams (mg), SC, once weekly from week 26 through week 52
  Metformin: at least 1500 milligrams per day (mg/day), oral, for 52 weeks
  Pioglitazone: at least 30 mg/day, oral, for 52 weeks
  All events were treatment emergent during the LY2189265 treatment period.
Arm/Group | 0.75 mg LY2189265 (Baseline Through 26 Weeks) | 1.5 mg LY2189265 (Baseline Through 26 Weeks) | Exenatide (Baseline Through 26 Weeks) | Placebo (Baseline Through 26 Weeks) | 0.75 mg LY2189265 (Baseline Through 56 Weeks) | 1.5 mg LY2189265 (Baseline Through 56 Weeks) | Exenatide (Baseline Through 56 Weeks) | Placebo/0.75 mg LY2189265 (26 Weeks Through 56 Weeks) | Placebo/1.5 mg LY2189265 (26 Weeks Through 56 Weeks)
Serious Adverse Events (participants affected / at risk) | 15/280 | 12/279 | 15/278 | 12/141 | 22/280 | 18/279 | 27/278 | 6/62 | 9/62
Other Adverse Events (participants affected / at risk) | 194/280 | 215/279 | 196/278 | 103/141 | 218/280 | 228/279 | 223/278 | 47/62 | 55/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 0.75 mg LY2189265 (Baseline Through 26 Weeks) (N=280) | 1.5 mg LY2189265 (Baseline Through 26 Weeks) (N=279) | Exenatide (Baseline Through 26 Weeks) (N=278) | Placebo (Baseline Through 26 Weeks) (N=141) | 0.75 mg LY2189265 (Baseline Through 56 Weeks) (N=280) | 1.5 mg LY2189265 (Baseline Through 56 Weeks) (N=279) | Exenatide (Baseline Through 56 Weeks) (N=278) | Placebo/0.75 mg LY2189265 (26 Weeks Through 56 Weeks) (N=62) | Placebo/1.5 mg LY2189265 (26 Weeks Through 56 Weeks) (N=62)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Event resulted in one death in the 1.5 mg LY2189265 group
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal sphincter insufficiency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Thrombosis in device (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Human anaplasmosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis syndrome (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/168 (0) | 0/163 (0) | 0/157 (0) | 1/83 (1) | 0/168 (0) | 0/163 (0) | 0/157 (0) | 0/36 (0) | 0/35 (0)
Prostate cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/168 (0) | 0/163 (0) | 0/157 (0) | 0/83 (0) | 1/168 (1) | 0/163 (0) | 0/157 (0) | 0/36 (0) | 0/35 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impaired self-care (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder perforation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0/112 (0) | 1/116 (1) | 0/121 (0) | 0/58 (0) | 0/112 (0) | 1/116 (1) | 0/121 (0) | 0/26 (0) | 0/27 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rehabilitation therapy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.75 mg LY2189265 (Baseline Through 26 Weeks) (N=280) | 1.5 mg LY2189265 (Baseline Through 26 Weeks) (N=279) | Exenatide (Baseline Through 26 Weeks) (N=278) | Placebo (Baseline Through 26 Weeks) (N=141) | 0.75 mg LY2189265 (Baseline Through 56 Weeks) (N=280) | 1.5 mg LY2189265 (Baseline Through 56 Weeks) (N=279) | Exenatide (Baseline Through 56 Weeks) (N=278) | Placebo/0.75 mg LY2189265 (26 Weeks Through 56 Weeks) (N=62) | Placebo/1.5 mg LY2189265 (26 Weeks Through 56 Weeks) (N=62)
Constipation (Gastrointestinal disorders) | 5 (6) | 12 (15) | 5 (6) | 2 (2) | 5 (6) | 16 (19) | 5 (6) | 2 (2) | 4 (6)
Diarrhoea (Gastrointestinal disorders) | 22 (42) | 31 (55) | 16 (22) | 8 (12) | 26 (47) | 37 (67) | 22 (38) | 5 (14) | 8 (8)
Dyspepsia (Gastrointestinal disorders) | 5 (6) | 22 (36) | 19 (19) | 4 (4) | 6 (7) | 23 (37) | 21 (21) | 0 (0) | 6 (9)
Flatulence (Gastrointestinal disorders) | 3 (4) | 14 (15) | 6 (7) | 3 (3) | 3 (4) | 16 (17) | 7 (8) | 0 (0) | 3 (4)
Nausea (Gastrointestinal disorders) | 45 (60) | 78 (108) | 71 (86) | 8 (8) | 47 (64) | 82 (114) | 77 (101) | 6 (6) | 15 (17)
Vomiting (Gastrointestinal disorders) | 17 (29) | 47 (67) | 30 (40) | 2 (2) | 17 (29) | 48 (68) | 34 (52) | 3 (5) | 5 (5)
Fatigue (General disorders) | 12 (16) | 10 (11) | 21 (21) | 2 (3) | 13 (17) | 13 (14) | 22 (23) | 3 (5) | 2 (2)
Oedema peripheral (General disorders) | 13 (13) | 3 (3) | 11 (12) | 7 (7) | 15 (16) | 8 (8) | 17 (18) | 9 (10) | 3 (3)
Influenza (Infections and infestations) | 8 (8) | 5 (5) | 7 (8) | 4 (4) | 12 (12) | 12 (13) | 14 (16) | 4 (5) | 3 (3)
Nasopharyngitis (Infections and infestations) | 23 (26) | 18 (19) | 12 (12) | 8 (8) | 26 (33) | 28 (31) | 16 (17) | 5 (6) | 2 (2)
Sinusitis (Infections and infestations) | 6 (6) | 5 (5) | 10 (10) | 2 (2) | 9 (11) | 12 (15) | 16 (16) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 14 (17) | 12 (13) | 12 (14) | 6 (8) | 25 (31) | 16 (18) | 20 (29) | 5 (6) | 4 (5)
Urinary tract infection (Infections and infestations) | 8 (8) | 11 (11) | 6 (6) | 4 (4) | 13 (15) | 16 (18) | 14 (14) | 2 (2) | 5 (5)
Lipase increased (Investigations) | 3 (3) | 7 (8) | 5 (6) | 4 (4) | 6 (6) | 9 (11) | 9 (11) | 4 (5) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 14 (14) | 22 (23) | 8 (8) | 3 (3) | 15 (16) | 23 (24) | 9 (9) | 2 (3) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10) | 8 (9) | 9 (12) | 3 (3) | 17 (18) | 12 (13) | 13 (19) | 3 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 11 (11) | 8 (9) | 9 (9) | 14 (16) | 15 (16) | 12 (14) | 4 (4) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (9) | 6 (6) | 8 (8) | 6 (7) | 13 (14) | 12 (12) | 15 (17) | 3 (4) | 4 (4)
Dizziness (Nervous system disorders) | 8 (9) | 15 (19) | 18 (23) | 2 (2) | 10 (11) | 19 (24) | 21 (30) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 9 (10) | 20 (26) | 24 (27) | 8 (9) | 14 (15) | 26 (36) | 25 (31) | 5 (6) | 6 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | 3 (3) | 7 (7) | 7 (8) | 7 (9) | 3 (3) | 4 (4) | 5 (5)
Hypertension (Vascular disorders) | 6 (6) | 7 (7) | 3 (3) | 6 (6) | 7 (7) | 8 (8) | 6 (6) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days